CLINICAL TRIAL: NCT05977049
Title: Psychosocial Support for Patients With Takotsubo Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-04025981
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Takotsubo Cardiomyopathy
Keywords: Takotsubo; Cardiomyopathy; Takotsubo Syndrome
MeSH Terms: conditions — Takotsubo Cardiomyopathy; Cardiomyopathies

STUDY DESIGN:
Intervention Model Description: All subjects will be placed in a virtual Takotsubo Support Group once enrolled in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Takotsubo Support Group (Other): Participants diagnosed with Takotsubo Syndrome will be enrolled into the study.
  Interventions: Behavioral: Takotsubo Support Group

INTERVENTIONS:
Behavioral: Takotsubo Support Group — Participants will undergo virtual group therapy/education. Participants will meet once every other week (at minimum), for 1 - 1.5 hours (on average). The frequency and/or length of the support group sessions may be adjusted according to participants' needs.

SUMMARY:
The study hypothesis is that participants enrolled in a virtual Takotsubo support group will have significantly less anxiety at one year.

DETAILED DESCRIPTION:
Takotsubo cardiomyopathy, sometimes termed Takotsubo syndrome and "broken heart syndrome," typically presents with symptoms remarkably similar to acute myocardial infarction (MI; heart attack): debilitating chest pain, shortness of breath, and a feeling of doom, among others. Takotsubo was first identified in 1990 in Japan. Most cases occur in older women. During the acute phase, the heart spontaneously undergoes "apical ballooning," changing shape to resemble a "takotsubo," a Japanese octopus trap. In approximately two-thirds of cases, Takotsubo is precipitated by an intense emotional or physical "trigger." Typically, the heart spontaneously reverts to its previous shape within about a month. Initially, it was thought that recurrence was rare. However, more recently, recurrences have been reported in 3-15% of cases. Many patients experience a variety of debilitating cardiac and psychological symptoms long after the initial presentation. There is no known way to prevent a recurrent event and patients are typically anxious about the possibility.

Since its inception as a diagnosis, one of the hallmarks of Takotsubo has been the absence of coronary artery plaque. In a surprising finding from 2019, a study of more than 1,000 Takotsubo patients undergoing coronary angiography reported that approximately 1/3 of patients had clinically significant plaque in their coronary arteries; 1/3 had evidence of sub-clinical atherosclerosis; and 1/3 had "clean coronaries," with no observable plaque. Hence, much needs to be learned about this syndrome that may affect as many as 5% of women who have been diagnosed with acute MI. Takotsubo is typically an emotionally challenging and life altering event. Strategies for primary and secondary prevention of coronary artery disease will be discussed in the virtual group sessions.

Currently, there is no specialized intervention for patients diagnosed with Takotsubo Syndrome at Weill Cornell Medical Center, either in hospital or after discharge.

ELIGIBILITY:
Inclusion Criteria:

- All patients with documented diagnosis of Takotsubo Syndrome greater than 18 years old.

Exclusion Criteria:

* Patients with a diagnosis of Takotsubo Syndrome already undergoing Psychotherapy or those who choose not to participate.
* Vulnerable populations such as prisoners, non-English speaking subjects, pregnant women, and subjects unable to provide written informed consent will not be included in this research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety level as measured by the STAI. | Baseline, One year
  State Trait Anxiety Inventory (STAI):
  Score of 20-39 = Low Anxiety; Score of 40-59 = Moderate Anxiety; Score of 60 - 80 = High Anxiety

SECONDARY OUTCOMES:
Changes in depression as measured by the PHQ-8. | Baseline, One year
  Patient Health Questionnaire depression scale (PHQ-8):
  Score of 0-2 = No Depression; Score of 3-5 = Mild Depression; Score of 6-8 = Moderate Depression; Score of 9-12 = Severe Depression
Changes in quality of life as measured by the KCCQ. | Baseline, One year
  Kansas City Quality of Life Questionnaire (KCCQ):
  Score of 0-24 = Very poor to poor quality of life; Score of 25-49 = Poor to fair quality of life; Score of 50-74 = Fair to good quality of life; Score of 75-100 = Good to excellent quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Jim Cheung, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sato, H., et al. (1990) Takotsubo-type cardiomyopathy due to multivessel spasm. In: Kodama, K., Haze, K., Hon M, et al., Eds., Clinical Aspect of Myocardial Injury: From Ischemia to Heart Failure, Kagakuhyouronsha, Tpkyo, 56-64.
- [Background] Ghadri JR, Wittstein IS, Prasad A, Sharkey S, Dote K, Akashi YJ, Cammann VL, Crea F, Galiuto L, Desmet W, Yoshida T, Manfredini R, Eitel I, Kosuge M, Nef HM, Deshmukh A, Lerman A, Bossone E, Citro R, Ueyama T, Corrado D, Kurisu S, Ruschitzka F, Winchester D, Lyon AR, Omerovic E, Bax JJ, Meimoun P, Tarantini G, Rihal C, Y-Hassan S, Migliore F, Horowitz JD, Shimokawa H, Luscher TF, Templin C. International Expert Consensus Document on Takotsubo Syndrome (Part I): Clinical Characteristics, Diagnostic Criteria, and Pathophysiology. Eur Heart J. 2018 Jun 7;39(22):2032-2046. doi: 10.1093/eurheartj/ehy076. PMID 29850871
- [Background] Napp LC, Cammann VL, Jaguszewski M, Szawan KA, Wischnewsky M, Gili S, Knorr M, Heiner S, Citro R, Bossone E, D'Ascenzo F, Neuhaus M, Franke J, Sorici-Barb I, Noutsias M, Burgdorf C, Koenig W, Kherad B, Sarcon A, Rajan L, Michels G, Pfister R, Cuneo A, Jacobshagen C, Karakas M, Pott A, Meyer P, Arroja JD, Banning A, Cuculi F, Kobza R, Fischer TA, Vasankari T, Airaksinen KEJ, Hauck C, Paolini C, Bilato C, Imori Y, Kato K, Kobayashi Y, Opolski G, Budnik M, Dworakowski R, MacCarthy P, Kaiser C, Osswald S, Galiuto L, Dichtl W, Chan C, Bridgman P, Beug D, Delmas C, Lairez O, El-Battrawy I, Akin I, Gilyarova E, Shilova A, Gilyarov M, Horowitz JD, Polednikova K, Tousek P, Widimsky P, Winchester DE, Galuszka J, Ukena C, Poglajen G, Carrilho-Ferreira P, Di Mario C, Prasad A, Rihal CS, Schulze PC, Bianco M, Crea F, Borggrefe M, Maier LS, Pinto FJ, Braun-Dullaeus RC, Rottbauer W, Katus HA, Hasenfuss G, Tschope C, Pieske BM, Thiele H, Schunkert H, Bohm M, Felix SB, Munzel T, Bax JJ, Bauersachs J, Braunwald E, Luscher TF, Ruschitzka F, Ghadri JR, Templin C. Coexistence and outcome of coronary artery disease in Takotsubo syndrome. Eur Heart J. 2020 Sep 7;41(34):3255-3268. doi: 10.1093/eurheartj/ehaa210. PMID 32484517